CLINICAL TRIAL: NCT00078988
Title: A Phase III Randomized Trial for the Treatment of Pediatric High Grade Gliomas at First Recurrence With a Single High Dose Chemotherapy and Autologous Stem Cell Transplant Versus Three Courses of Intermediate Dose Chemotherapy With Peripheral Blood Stem Cell (PBSC) Support
Brief Title: High-Dose Chemotherapy Plus Autologous Stem Cell Transplantation Compared With Intermediate-Dose Chemotherapy Plus Autologous Stem Cell Transplantation With or Without Isotretinoin in Treating Young Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0231; COG-ACNS0231 (Other: Children's Oncology Group); CDR0000353207 (Other: NCI); NCI-2012-02578 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA098543 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: childhood high-grade cerebral astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Astrocytoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Etoposide; etoposide phosphate; Isotretinoin; Thiotepa; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (high-dose chemotherapy and ASCR) (Experimental): Patients receive high-dose chemotherapy comprising carboplatin IV over 4 hours on days -8 to -6; thiotepa IV over 3 hours and etoposide IV over 3 hours on days -5 to -3; and filgrastim (G-CSF) IV or SC once daily beginning on day 1 and continuing until blood counts recover. Autologous PBSC or bone marrow are reinfused on day 0.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: isotretinoin; Drug: thiotepa; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation
- Arm II (intermediate-dose chemotherapy and ASCR) (Experimental): Patients receive intermediate-dose chemotherapy comprising carboplatin IV over 4 hours and thiotepa IV over 3 hours on days 1-2 and G-CSF IV or SC once daily beginning on day 4 and continuing until blood counts recover. Autologous PBSC or bone marrow are reinfused on day 3. Treatment repeats every 28 days for a total of 3 courses.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: thiotepa; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation
- Arm III (isotretinoin) (Experimental): Patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for a total of 6 courses.
  Interventions: Drug: isotretinoin
- Arm IV (no isotretinoin) (No Intervention): Patients do not receive maintenance therapy.

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC 614629
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm II (intermediate-dose chemotherapy and ASCR)
Drug: carboplatin — Given IV
  Other Names: Paraplain; CBDCA; NSC #241240
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm II (intermediate-dose chemotherapy and ASCR)
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
  Arms: Arm I (high-dose chemotherapy and ASCR)
Drug: isotretinoin — Given IV
  Other Names: 13-cis-retinoic acid; RO-43; 780; Accutane; NSC#329481
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm III (isotretinoin)
Drug: thiotepa — Given IV
  Other Names: Tespa; Thiophosphamide; Triethylenethiophosphoramide Tspa; WR-45312; NSC#6396
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm II (intermediate-dose chemotherapy and ASCR)
Procedure: autologous bone marrow transplantation — Peripheral blood stem cells or bone marrow will be reinfused about 72 hours following completion of the last dose of chemotherapy (Day 0)
  Other Names: Stem Cell Reinfusion
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm II (intermediate-dose chemotherapy and ASCR)
Procedure: peripheral blood stem cell transplantation — Filgrastim is to be given daily in the afternoon for 4 days prior to the first harvest and continued until the completion of the daily harvests. The daily PBSC harvesting should be started prior to the fifth dose of filgrastim.
  Other Names: Peripheral Stem Cell Collection
  Arms: Arm I (high-dose chemotherapy and ASCR); Arm II (intermediate-dose chemotherapy and ASCR)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, thiotepa, and etoposide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Isotretinoin may be effective in preventing recurrence of glioma. It is not yet known which regimen of chemotherapy plus autologous stem cell transplantation with or without isotretinoin is more effective in treating recurrent high-grade glioma.

PURPOSE: This randomized phase III trial is studying high-dose chemotherapy or intermediate-dose chemotherapy followed by autologous stem cell transplantation to see how well it works compared to high-dose chemotherapy or intermediate-dose chemotherapy followed by autologous stem cell transplantation and isotretinoin in treating young patients with recurrent high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival and overall survival of pediatric patients with recurrent high-grade gliomas treated with a single course of high-dose carboplatin, etoposide, and thiotepa and autologous stem cell transplantation vs multiple courses of intermediate-dose carboplatin and thiotepa and autologous stem cell transplantation with or without isotretinoin.
* Compare the number of hospital days and time to engraftment in patients treated with these regimens.
* Compare the toxic death rate in patients treated with these regimens.
* Compare the tolerability of isotretinoin in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to pathologic diagnosis (glioblastoma multiforme vs anaplastic astrocytoma vs other high-grade glioma).

* Chemotherapy and autologous stem cell reinfusion (ASCR): Patients are randomized to 1 of 2 treatment arms.

  * Arm I (high-dose chemotherapy and ASCR): Patients receive high-dose chemotherapy comprising carboplatin IV over 4 hours on days -8 to -6; thiotepa IV over 3 hours and etoposide IV over 3 hours on days -5 to -3; and filgrastim (G-CSF) IV or subcutaneously (SC) once daily beginning on day 1 and continuing until blood counts recover. Autologous peripheral blood stem cells (PBSC) or bone marrow are reinfused on day 0.
  * Arm II (intermediate-dose chemotherapy and ASCR): Patients receive intermediate-dose chemotherapy comprising carboplatin IV over 4 hours and thiotepa IV over 3 hours on days 1-2 and G-CSF IV or SC once daily beginning on day 4 and continuing until blood counts recover. Autologous PBSC or bone marrow are reinfused on day 3. Treatment repeats every 28 days for a total of 3 courses.
* Maintenance therapy: After recovery from chemotherapy (approximately day 30 post-transplantation), all patients are further randomized to 1 of 2 maintenance arms.

  * Arm I: Patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for a total of 6 courses.
  * Arm II: Patients do not receive maintenance therapy. In all arms, treatment continues in the absence of disease progression.

Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 80-150 patients (40-75 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following high-grade gliomas:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Gliosarcoma
* Disease in first relapse
* No primary brainstem or spinal cord gliomas
* No secondary glioblastomas arising after prior treatment for a non-glial tumor
* Prior local radiotherapy of 5,000-6,000 cGy required
* Less than 1.5 cm of residual gadolinium-enhancing tumor in maximal cross-sectional diameter by MRI
* No metastatic tumor by spinal MRI

PATIENT CHARACTERISTICS:

Age

* Under 21 at diagnosis

Performance status

* Lansky 50-100% OR
* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 500/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN

Renal

* Glomerular filtration rate ≥ 60 mL/min AND/OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* Shortening fraction ≥ 27% by echocardiogram OR
* Ejection fraction ≥ 50% by MUGA

Pulmonary

* No dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No prior thiotepa
* No prior myeloablative chemotherapy

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* See Disease Characteristics
* More than 8 weeks since prior radiotherapy
* No prior craniospinal radiotherapy

Surgery

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2004-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Event-free survival | om study entry to disease progression, disease relapse, occurrence of a second malignant neoplasm, or death from any cause. assessed up to 4 years
  The primary endpoint for the evaluation of treatment efficacy will be event-free survival (EFS)
Toxic death attributable to complications of treatment in the absence of tumor progression as assessed by NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0 | Up to 4 years after completion of study treatment
  Toxic death will be monitored separately in each of the two chemotherapy groups

SECONDARY OUTCOMES:
Overall survival (OS) | ondary e ndpoints include overall survival (OS), which is defined as the time from study entry to death from any cause assessed up to 4 years
  Secondary endpoints include overall survival (OS), which is defined as the time from study entry to death from any cause, assessed up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Khatib, MD, Study Chair — Nicklaus Children's Hospital f/k/a Miami Children's Hospital; Sharon L. Gardner, MD, Study Chair — NYU Langone Health
Locations (59):
- United States (52):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - University of California Davis Cancer Center, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (6):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec